CLINICAL TRIAL: NCT03500783
Title: Nitric Oxide-mediated Cardioprotection During Cardiac Surgery With Cardiopulmonary Bypass
Acronym: NOinCPB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Nikolay Kamenshchikov, Principal Investigator, Physician Anesthesiologist, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NOinCPB
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass; Cardiopulmonary Bypass; Nitric Oxide; Reperfusion Injury, Myocardial
Keywords: Cardioprotection; Ischemia-reperfusion injury; Nitric oxide; Cardiopulmonary bypass; Coronary artery bypass grafting
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Reperfusion Injury; Reperfusion Injury | interventions — Nitric Oxide; Cardiopulmonary Bypass

STUDY DESIGN:
Intervention Model Description: Single-center prospective, randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Trial participants, data analysts, and report writers are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide (Experimental): Patients of this group receive treatment with exogenous gaseous nitric oxide supplied directly to the oxygenator in the cardiopulmonary bypass circuit during coronary artery bypass grafting for coronary artery disease.
  Interventions: Drug: Nitric Oxide
- Standard CPB (Placebo Comparator): Patients of this group receive sham-treatment without supplying nitric oxide to the cardiopulmonary bypass circuit during coronary artery bypass grafting for coronary artery disease. Considering dilution of nitric oxide at a high ratio of 1 to 25,000 in the gas mixture of the cardiopulmonary bypass circuit (CPB), no addition of any inert gas to the CPB circuit is required in sham-treatment group.
  Interventions: Other: Standard CPB

INTERVENTIONS:
Drug: Nitric Oxide — 40 ppm of exogenous gaseous nitric oxide is supplied directly to the oxygenator in the cardiopulmonary bypass circuit during coronary artery bypass grafting.
  Arms: Nitric Oxide
Other: Standard CPB — Standard protocol of delivery of air gas mixture to the cardiopulmonary bypass circuit
  Other Names: Cardiopulmonary bypass
  Arms: Standard CPB

SUMMARY:
This prospective randomized study elucidates the effects of exogenous nitric oxide delivered to the extracorporeal circulation circuit for cardioprotection against ischemia-reperfusion injury during coronary artery bypass graft surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of exogenous nitric oxide (NO) delivered to the extracorporeal circulation circuit for cardioprotection against ischemia-reperfusion injury during coronary artery bypass graft surgery (CABG) with cardiopulmonary bypass (CPB). A total of 60 patients with ischemic heart disease referred for CABG with CPB are included in prospective randomized study. Patients are randomized to receive standard treatment or surgery based on modified CPB protocol. According to modified protocol, 40-ppm NO is supplied to the CPB circuit during CABG. The primary endpoints are changes in cardiac troponin I (cTnI) levels at 6, 24, and 48 hours after surgery compared with baseline. The secondary end points are the changes in the levels of creatine kinase-muscle/brain (CK-MB) compared with baseline and vasoactive inotropic score (VIS) at 6, 24, and 48 hours. NO supplied to the CPB circuit exertes cardioprotective effect. Changes in cTnI, CK-MB, and VIS are considered indictors of the presence or absence of cardioprotective action of NO supplied to the CPB circuit.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease requiring coronary artery bypass grafting with the cardiopulmonary bypass.

Exclusion Criteria:

* Non-elective surgery, age over 70 years, left ventricular ejection fraction less than 35%, history of myocardial infarction within three months prior to surgery, chronic atrial fibrillation, diabetes mellitus, and the elevated levels of cardiac specific markers within 12 h prior to the intervention.

Ages: 56 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Cardiac troponin I change measure (cTnI) | 48 hours (with intermediate measurements at 6 and 24 hours)
  Changes in the plasma level of cTnI (ng/mL) relative to the baseline value are measured at 6, 24, and 48 hours after surgery.

SECONDARY OUTCOMES:
Creatine kinase-muscle/brain change measure (CK-MB) | 48 hours (with intermediate measurements at 6 and 24 hours)
  Changes in the plasma level of CK-MB (U/L) relative to the baseline value are measured at 6, 24, and 48 hours after surgery.
Vasoactive inotropic score measure (VIS) | 48 hours (with intermediate measurements at 6 and 24 hours)
  Vasoactive inotropic score (VIS) is assessed at 6, 24, and 48 hours after surgery. VIS is calculated as follows: (dobutamine μg/kg/min × 1 + dopamine μg/kg/min × 1 + milrinone μg/kg/min × 10) + 100 × (adrenalin μg/kg/min + noradrenaline μg/kg/min + vasopressin μg/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Popov, MD, Study Director — Tomsk NRMC

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.